Version: 01 Version date: September 9, 2024

informed consent

( intervention study )

Name of research project: Application of PDCA teaching mode in emergency resident physician

tracheal intubation teaching and training

Version number of informed consent: 1.0 September 9, 2024

Research institution: Panyu Central Hospital affiliated to Guangzhou Medical University

Lead Investigator:

By Mr./Ms.:

You will be invited to participate in a study titled "Application of the PDCA Teaching Model in Emergency Department Resident Tracheal Intubation Training". This informed consent document provides detailed information to help you decide whether to join this program. Please

read it carefully. If you have any questions, please contact the investigator responsible for this

research, and we will provide comprehensive explanations.

Your participation in this study is completely voluntary. This study has been reviewed by the

Medical Ethics Committee of Panyu Central Hospital affiliated to Guangzhou Medical University.

1. Research Background

Tracheal intubation is a vital lifesaving technique in emergency care, recognized as one of

the most widely used, effective, and efficient methods for airway management. As an essential

skill for emergency physicians, mastering this procedure significantly improves treatment success

rates for critically ill patients. This underscores the critical importance of providing tracheal

intubation training to emergency department practitioners.

2. Research Objectives

This study aims to explore the application effect of PDCA model in emergency department

rotation and resident intubation teaching training, and provide reference for related teaching

activity reform.

3. The time of study and the number of participants

This study will be conducted in the emergency department and is expected to include 100

1

qualified subjects. The study is expected to last one month.

### 4. Research process

If you participate in this study, after signing the informed consent form, we will use the PDCA mode of teaching method. During the research process, we need to collect your major, age, working age, teaching satisfaction, theoretical and practical performance, success rate of tracheal intubation and other data.

## 5. Who should not participate in the study

If you have previously participated in a tracheal intubation training, you should not participate in this study:

### 6. Matters requiring your cooperation

In order to make this research smooth and successful, please cooperate with the following:

· Study according to the researcher's arrangement.

### 7. Risks and discomforts of participating in research

If you feel that the teaching method is not suitable for your study or causes any discomfort during this experiment, please report to the instructor in time and withdraw from this experiment.

# 8. Participate in research about possible benefits

You and society may benefit directly or indirectly from this research, including the possibility of improved learning and the potential for this research to inform teaching reforms.

#### 9. Alternative treatment options

In addition to participating in this study, you have the following options: Study using conventional teaching methods.

#### 10. Relevant costs of participation in the study

The research costs related to this project will be borne by the research group, and you will not need any money.

#### 11. Compensation

not have .

#### 12. Study of medical and compensation for related injuries

If any damage related to this study is found to be liable by an authoritative institution in accordance with national laws and regulations, the researcher will assume the liability and make corresponding compensation in accordance with Chinese laws.

#### 13. Right to refuse or withdraw from the study

You may choose not to participate in this study or, at any time, notify the investigator of your request to withdraw from the study. The data collected about you prior to this will not be included in the results of the study and will not affect your treatment or rights.

If you do not follow the research plan, or for any reason you want to withdraw from the project, you may ask your supervisor.

## 14. Privacy and confidentiality issues

If you decide to participate in this study, your personal information during the trial will be kept confidential. Your identity details will not be disclosed to anyone outside the research team unless you explicitly authorize it. All participants and sponsors are required to maintain strict confidentiality regarding your identity. Your medical records will be stored in a locked file cabinet exclusively accessible to researchers. To ensure compliance with regulations, government authorities or ethics review committee members may access your personal data at the research facility following standard approval procedures. When the study results are published, no personally identifiable information about you will be disclosed.

#### How to get help in research

You can learn about the information and research progress related to this study at any time. If you have questions related to this study, or if you experience any discomfort or injury during the study, or if you have questions about the rights and interests of participants in this study, you can contact the relevant person by phone. Contact person:\_\_\_\_\_\_ contact number : \_\_\_\_\_

For equity related issues, please contact the Hospital Ethics Committee at 020-34858239.

If you fully understand the contents of this research project and agree to participate in this study, you will sign this INFORMED consent form in duplicate, with one copy retained by the investigator and one copy by the subject or the client.

# Informed consent statement of the subject

I have read and fully understood the above introduction to this study, and have had the opportunity to discuss and ask questions about this study with the doctor. All my questions have been answered satisfactorily.

I understand the risks and benefits of participating in this study. I understand that participation is voluntary.

Version: 01 Version date: September 9, 2024 Version: 01 Version date: September 9, 2024 Subject signed Signature Date: Year Month Day Minute Contact number: Signature Date: Year Month Day Minute Contact number:\_\_\_\_ Signature of impartial witness (if necessary)\_\_\_\_ Signature Date: Year Month Day Minute Contact number: Signature Date: Year Month Day Minute Contact number:\_\_\_\_\_ Guardian's signature (if necessary)\_\_\_\_\_ Signature Date: Year Month Day Minute Contact number: Signature Date: Year Month Day Minute Contact number: Study authors declare I confirm that the patient has been informed of the details of this study, including their rights and possible benefits and risks, and that questions raised by the subject have been addressed in detail. The study was signed by the researcher\_\_\_\_\_

(Note: If the subject is illiterate, a fair witness signature is required; if the subject is

Signature Date:

Signature Date: Year Month Day Minute Contact number:

Year Month Day Minute Contact number:

incompetent, a guardian signature is required)